CLINICAL TRIAL: NCT06393855
Title: Base Curves of Bandage Contact Lenses and Their Effects on Post Transepithelial Photorefractive Keratectomy (Trans-PRK) Vision and Pain： A Prospective Randomized Clinical Trial
Brief Title: Base Curves of Bandage Contact Lenses and Their Effects on Post Trans-PRK Vision and Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dongyang People's Hospital (Other)
Responsible Party: Principal Investigator, Gengmin Tong, Doctor, Dongyang People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCLTPRK
Record Dates: First submitted 2024-04-22; First posted 2024-05-01 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Myopia
Keywords: Transepithelial photorefractive keratectomy; High Myopia; bandage contact lenses
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- contact lens with 8.4-mm base curve in right eye (Experimental): A contact lens placed on the cornea after the single-step Trans-PRK，with an 8.4-mm base curve in right eye and one with an 8.8-mm base curve in the left eye
  Interventions: Procedure: single-step Trans-PRK; Behavioral: Placing a bandage contact lens on the cornea, with an 8.4-mm base curve in right eye and one with an 8.8-mm base curve in the left eye.
- contact lens with 8.8-mm base curve in right eye (Experimental): A contact lens placed on the cornea after the single-step Trans-PRK，with an 8.8-mm base curve in right eye and one with an 8.4-mm base curve in the left eye
  Interventions: Procedure: single-step Trans-PRK; Behavioral: Placing a bandage contact lens on the cornea,A contact lens placed on the cornea, with an 8.8-mm base curve in right eye and one with an 8.4-mm base curve in the left eye.

INTERVENTIONS:
Procedure: single-step Trans-PRK — Both eyes were treated consecutively in each patient by single-step Trans-PRK performed by SCHWIND Amaris 500 S excimer laser platform (SCHWIND eye-tech-solutions GmbH, Kleinostheim, Germany). Topical Proparacaine Hydrochloride Eye Drops 0.5% (Alcaine, Alcon, Fort Worth, TX, USA) were used to anesthetize the eyes, and use povidone-iodine to disinfect the eyelid skin. After a lid speculum had been inserted, and the other eye was blocked. Epithelial and stromal ablations were performed using a single continuous laser shooting session on an excimer laser platform. After the appeals step, Mitomycin C 0.02 % was applied to the stromal surface for 20 s, then rinse with cold salt water.
Behavioral: Placing a bandage contact lens on the cornea, with an 8.4-mm base curve in right eye and one with an 8.8-mm base curve in the left eye. — After surgery. A contact lens placed on the cornea, with an 8.4-mm base curve in right eye and one with an 8.8-mm base curve in the left eye.
  Arms: contact lens with 8.4-mm base curve in right eye
Behavioral: Placing a bandage contact lens on the cornea,A contact lens placed on the cornea, with an 8.8-mm base curve in right eye and one with an 8.4-mm base curve in the left eye. — After surgery. A contact lens placed on the cornea, with an 8.8-mm base curve in right eye and one with an 8.4-mm base curve in the left eye.
  Arms: contact lens with 8.8-mm base curve in right eye

SUMMARY:
The objective of this study was to investigate the impact of employing bandage contact lenses with a base curve of 8.4 mm versus 8.8 mm on visual recovery following Trans-PRK in patients characterized by steep corneas and high myopia.

DETAILED DESCRIPTION:
Comparing two kind of bandage lenses in the contralateral eyes of the same individual following Trans-PRK may enable the derivation of reliable conclusions regarding the optimal choice for bandage lenses after Trans-PRK.

ELIGIBILITY:
Inclusion Criteria:

Spherical equivalent refractive error between -6.00 and -8.00 D in either eye.

Astigmatism of no more than 2.0 D in either eye.

Best spectacle-corrected visual acuity (BCVA) according to the logarithm of the Minimum angle of resolution (logMAR) scale of 0 or better in both eyes.

Willing and able to participate in all required activities of the study.

Exclusion Criteria:

Diabetes mellitus.

Systemic connective tissue disease.

Cardiovascular disease, epilepsy.

Eyelid abnormalities.

Corneal disease.

Glaucoma.

A history of ocular disease.

Noncompliance with measurement at enrollment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Early postoperative uncorrected visual acuity | 14 days
  All visual acuity measurements were performed using a standard logarithmic eye chart

SECONDARY OUTCOMES:
re-epithelialization after Trans-PRK | 1 week
  A ophthalmologist will examine the corneal epithelium in all eyes. The assessment of corneal epithelial defects involves measuring the horizontal and vertical diameters using a slit lamp beam with a ruler. The extent of corneal epithelial defects is determined by calculating the area of the ellipse (S=πa×b).
postoperative pain score after Trans-PRK | 2 weeks
  Patients will be asked to complete a pain questionnaire at postoperative 0, 2, 12 hours and 1, 4, 7, 14 days. A visual analog scale (VAS) was employed to assess the severity of pain in each eye. The scores are defined as follows: 0 points: no pain; 1-3 points: mild pain, does not affect work and life; 4-6 points: moderate pain, affects work, does not affect life; 7-10 points: severe pain, affects both work and life
spherical equivalent after Trans-PRK | 1 week
  Optometry is performed using a computerized optometre. The spherical equivalent (SE) was calculated using the formula DS+DC/2, where DS denotes the diopter sphere and DC denotes the diopter cylinder.

CONTACTS AND LOCATIONS:
Overall Officials: Guangjin Zhao, Study Director — Dongyang People's Hospital
Locations (1):
- Dongyang People's Hospital, Dongyang, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tong G, Jin Y, Zhou H, Jin Y. Base curves of bandage contact lenses and their effects on post Trans-PRK vision and pain: the study protocol for a randomized clinical trial. Trials. 2025 Sep 25;26(1):357. doi: 10.1186/s13063-025-09115-y. PMID 40999507